CLINICAL TRIAL: NCT03035721
Title: Clinical Evaluation of a Low Protein Content Formula Fed to Full Term Healthy Infants in the First Months of Life: a Randomized Controlled Trial
Brief Title: Clinical Evaluation of a Low Protein Content Formula in the First Months of Life: a RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: Humana Co.Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Low protein formula_RCT
Record Dates: First submitted 2017-01-17; First posted 2017-01-30 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-01

CONDITIONS: Safety Issues; Infant Nutrition Disorders
Keywords: Full term healthy infants; Low protein content formula; Safety; Growth; Body composition
MeSH Terms: conditions — Infant Nutrition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Anthropometric and body composition measurements were performed by three medical investigators who were blinded to allocated treatment.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low protein formula group (Experimental): Full term healthy infants randomized to receive a low protein formula for the first 4 months of life
  Interventions: Dietary Supplement: Low protein formula
- Standard protein formula group (Active Comparator): Full term healthy infants randomized to receive a standard protein formula for the first 4 months of life
  Interventions: Dietary Supplement: Standard protein formula
- Breastfeeding group (No Intervention): Breastfed full term healthy infants

INTERVENTIONS:
Dietary Supplement: Low protein formula — Infants were enrolled to receive low protein formula (energy: 65 kcal/100 mL, protein: 1.2 g/100 mL, protein-to-energy ratio:1.9 g/100 kcal, carbohydrates: 8 g/100 mL, fat: 3.1 g/100 mL) for the firsts 4 months of life.
  Arms: Low protein formula group
Dietary Supplement: Standard protein formula — Infants were enrolled to receive standard protein formula (energy: 68 kcal/100 mL, protein: 1.7 g/100 mL, protein-to-energy ratio:2.5 g/100 kcal, carbohydrates: 7.1 g/100 mL, fat: 3.5 g/100 mL) for the firsts 4 months of life.
  Arms: Standard protein formula group

SUMMARY:
This study aimed to evaluate the tolerance and safety of a low-protein formula in healthy full-term infants by investigating effects on growth and gastrointestinal tolerance and by identifying any adverse effects.

DETAILED DESCRIPTION:
Infants were randomized to receive either a standard protein formula or a low-protein formula. The composition of the low-protein formula vs the standard formula was: energy (65 vs. 68 kcal/100 mL), protein (1.2 vs. 1.7 g/100 mL).

To investigate the safety of the low-protein formula without any bias, a 4-month intervention period was selected during which the infants were fed only formula.

Anthropometric parameters (weight, length, and head circumference) and body composition were assessed at enrollment, at 2 and 4 months' of age. Parents were asked to keep a diary on the occurrence of gastrointestinal symptoms or any other symptoms and were contacted every two weeks either by clinic visits or phone calls.

The reference group was constituted by a cohort of healthy, exclusively breastfed, full-term infants.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* singleton
* full-term infants (gestational age 37/0 to 41/6 weeks)
* birth weight adequate for gestational age (>p10 and <p90 for gestational age) according to the World Health Organization growth charts.

Exclusion Criteria:

* presence of congenital diseases
* presence of chromosomal abnormalities
* presence of conditions that could interfere with growth, such as brain, metabolic, cardiac and gastrointestinal diseases, perinatal infections.
* being born to mother affected by endocrine and/or metabolic diseases
* having a family history of allergic disease

Ages: 1 Day to 3 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2014-06; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Evaluate weight | enrollment, 2 months and 4 months
  Weight (g) of each baby was measured on an electronic scale accurate to 0.1 g (PEA POD Infant Body Composition System; Cosmed, Concord, CA, US). Body length was measured to the nearest 1 mm on a Harpenden neonatometer (Holtain, Crymych, UK).
Evaluate lenght | enrollment 2 months and 4 months
  Lenght (cm) of each baby was measured according standard procedures.
Evaluate head circumference | enrollment 2 months and 4 months
  Head circumference was measured to the nearest 1 mm using non-stretch measuring tape.
Evaluate body composition (fat mass and fat free mass) | enrollment, 2 months and 4 months
  Body composition [fat mass and fat free mass (g)]was assessed using an air-displacement plethysmography (PEA POD Infant Body Composition System; COSMED, Italy).
Evaluate weight increase | 2 months, 4 months
  Weight increase (g/day) was calculated as a change in body weight from weight at study enrollment divided by the time interval from enrolment to the assessment at 4 months Fat mass (g/day) and fat free mass (g/day) increases were also calculated.
Evaluate gastrointestinal tolerance | 2 months and 4 months
  Parents were asked to keep a diary on the occurrence of gastrointestinal symptoms or any other symptoms and were contacted every two weeks either by clinic visits or phone calls.
  The occurrence of spitting up, vomiting and colic, defined as intermittent attacks of abdominal pain when the baby screamed and drew up his/her legs but was well between episodes, was recorded. Colic was further classified as severe if the episodes were more than twice per day. Daily frequency of stool passage was also collected.
Evaluate occurence of adverse events | 2 months and 4 months
  Adverse events were assessed based on inquires to the parents and on their daily records.

SECONDARY OUTCOMES:
Evaluate body mass index (k/m2: weight/length2) | enrollment, 2 months and 4 months
  Body mass index [BMI: (Kg/m2)] was assessed for all infants enrolled at each study points.
Evaluate z-score | enrollment, 2 months and 4 months
  Z-scores values for age were then calculated using the z score calculator provided by WHO [WHO Anthro (version 3.2.2, January 2011)].

CONTACTS AND LOCATIONS:
Overall Officials: Paola Roggero, MD, Principal Investigator — NICU. Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico Milano, Milan, Italy, 20122
Locations (1):
- NICU, Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liotto N, Orsi A, Menis C, Piemontese P, Morlacchi L, Condello CC, Gianni ML, Roggero P, Mosca F. Clinical evaluation of two different protein content formulas fed to full-term healthy infants: a randomized controlled trial. BMC Pediatr. 2018 Feb 13;18(1):59. doi: 10.1186/s12887-018-1046-6. PMID 29439736